CLINICAL TRIAL: NCT00065156
Title: A Multicenter, Single-arm, Open-label Study of the Efficacy and Safety of Lenalidomide Monotherapy in Red Blood Cell Transfusion-dependent Subjects With Myelodysplastic Syndromes Associated With a Del(5q) Cytogenetic Abnormality.
Brief Title: Lenalidomide Safety/Efficacy in Myelodysplastic Syndromes (MDS) Associated With a Deletion (Del)(5q) Cytogenetic Abnormality
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-MDS-003; NCT00074126 (obsolete NCT alias)
Record Dates: First submitted 2003-07-17; First posted 2003-07-18 (Estimated); Results first posted 2010-06-09 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Myelodysplastic Syndromes
Keywords: MDS; CC-5013; Revlimid; Celgene
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenalidomide (Experimental)
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: lenalidomide — 10 mg orally once daily for 21 days out of a 28-day cycle (syncopated); subsequently amended (Amendment 1, dated 27 August 2003) to employ a continuous dosage regimen in which 10 mg was taken once daily for 28 day cycles (continuous). Subjects who initially began a syncopated regimen and who did not experience a dose-limiting adverse event were allowed to switch to the continuous regimen.
  Other Names: CC-5013

SUMMARY:
This study is a multicenter, single-arm, open-label study of oral lenalidomide monotherapy administered to red blood cell (RBC) transfusion-dependent subjects with low- or intermediate-1-risk Myelodysplastic Syndromes (MDS) associated with a del (5q31-33) cytogenetic abnormality. Screening procedures will take place within 28 days of the first day of lenalidomide treatment. Subjects will receive lenalidomide in 28-day cycles for up to 6 cycles, or until bone marrow disease progression or progression/relapse following erythroid hematologic improvement is documented. Study visits will occur every cycle (every 28 days) and laboratory monitoring to assess hematological parameters will occur every 14 days. Safety and efficacy assessments to be performed during the study are outlined in the Schedule of Study Assessments.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign an informed consent form
* Age 18 years or older at the time of signing the informed consent
* Must be able to adhere to the study visit schedule and other protocol requirements.
* Diagnosis of low or intermediate-1-risk International Prognostic Scoring System (IPSS) Myelodysplastic Syndromes (MDS) without an abnormality of chromosome 5 involving a deletion between bands q31 and q33.
* Red blood cell (RBC) transfusion-dependent anemia defined as having received greater than or equal to 2 units of RBCs within 8 weeks of the first day of study drug treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1 or 2.
* Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test within 7 days of starting study drug.
* Sexually active WCBP must agree to use adequate contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) while on study drug.
* WCBP must agree to have pregnancy tests every 4 weeks while on study drug.

Exclusion Criteria:

* Pregnant or lactating females
* Prior therapy with lenalidomide.
* An abnormality of chromosome 5 involving a deletion between bands q31 and q33.
* Lab Abnormality: Absolute neutrophil count (ANC) <500 cell/mm^3 (0.5*10^9/L)
* Lab Abnormality: Platelet count <50,000/mm^3 (50*10^9/L)
* Lab Abnormality: Serum creatinine >2.5 mg/dL (221 mmol/L)
* Lab Abnormality: Serum total bilirubin >2.0 mg/dL (34 mmol/L)
* Prior greater than or equal to grade 3 National Cancer Institute (NCI) Common Toxicity Criteria (CTC) allergic reaction/hypersensitivity to thalidomide.
* Clinically significant anemia due to factors such as iron, B12 or folate deficiencies, autoimmune or hereditary hemolysis or gastrointestinal bleeding
* If a marrow aspirate is not evaluable for storage iron, transferrin saturation must be > 20% and serum ferritin not less than 50 ng/mL
* Use of hematopoietic growth factors within 7 days of the first day of study drug treatment.
* Prior greater than or equal to grade 3 NCI CTC rash or any desquamation (blistering) while taking thalidomide.
* Chronic use (>2 weeks) of greater than physiologic doses of a corticosteroid agent (dose equivalent to >10 mg/day of prednisone) within 28 days of the first day of study drug treatment.
* Use of experimental or standard drugs (i.e. chemotherapeutic, immunosuppressive, and cytoprotective agents) for the treatment of MDS within 28 days of the first day of study drug treatment.
* Prior history of malignancy other than MDS (except basal cell or squamous cell carcinoma or carcinoma in situ of the cervix or breast) unless the subject has been free of disease for greater than or equal to 3 years.
* Use of any other experimental therapy within 28 days of the first day of study drug treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2003-06-01 (Actual); Primary Completion 2008-08-01 (Actual); Study Completion 2008-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan F List, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (32):
- United States (31):
  - Arizona Cancer Center, Scottsdale, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - Desert Hematology & Oncology Medical Group, Rancho Mirage, California
  - Stanford University Medical Center, Stanford, California
  - Mayo Clinic, Jacksonville, Florida
  - Cancer & Blood Disease Center, Lecanto, Florida
  - University of Miami Sylvester Comp Cancer Center, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Northwest Georgia Oncology - Wellstar Cancer Research, Marietta, Georgia
  - Rush-Presbyterian- St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Midwest Cancer Research Group, Skokie, Illinois
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University School of Medicine, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Hospital-Cornell, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Mt. Sinai Medical Center, New York, New York
  - University of Rochester- James P. Wilmot Cancer Center, Rochester, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Kaiser Permanente Northwest Region, Portland, Oregon
  - Western Pennsylvania Cancer Institute, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- St. Johannes Hospital, Duisburg, Germany

REFERENCES:
- [Background] Sekeres MA, Maciejewski JP, Giagounidis AA, Wride K, Knight R, Raza A, List AF. Relationship of treatment-related cytopenias and response to lenalidomide in patients with lower-risk myelodysplastic syndromes. J Clin Oncol. 2008 Dec 20;26(36):5943-9. doi: 10.1200/JCO.2007.15.5770. Epub 2008 Nov 17. PMID 19018091
- [Background] Prebet T, Cluzeau T, Park S, Sekeres MA, Germing U, Ades L, Platzbecker U, Gotze K, Vey N, Oliva E, Sugrue MM, Bally C, Kelaidi C, Al Ali N, Fenaux P, Gore SD, Komrokji R. Outcome of patients treated for myelodysplastic syndromes with 5q deletion after failure of lenalidomide therapy. Oncotarget. 2017 Jun 14;8(47):81926-81935. doi: 10.18632/oncotarget.18477. eCollection 2017 Oct 10. PMID 29137233
- [Result] List A, Dewald G, Bennett J, Giagounidis A, Raza A, Feldman E, Powell B, Greenberg P, Thomas D, Stone R, Reeder C, Wride K, Patin J, Schmidt M, Zeldis J, Knight R; Myelodysplastic Syndrome-003 Study Investigators. Lenalidomide in the myelodysplastic syndrome with chromosome 5q deletion. N Engl J Med. 2006 Oct 5;355(14):1456-65. doi: 10.1056/NEJMoa061292. PMID 17021321
- [Result] A.F. List, et.al. Results of the MDS-002 and -003 international phase II studies evaluating lenalidomide (CC-5013; Revlimid) in the treatment of transfusion-dependent (TD) patients with myelodysplastic syndrome (MDS). European Hematology Association 10th Conference June 2-5, 2005 Abstract #0772
- [Derived] Fenaux P, Giagounidis A, Selleslag D, Beyne-Rauzy O, Mittelman M, Muus P, Nimer SD, Hellstrom-Lindberg E, Powell BL, Guerci-Bresler A, Sekeres MA, Deeg HJ, Del Canizo C, Greenberg PL, Shammo JM, Skikne B, Yu X, List AF. Clinical characteristics and outcomes according to age in lenalidomide-treated patients with RBC transfusion-dependent lower-risk MDS and del(5q). J Hematol Oncol. 2017 Jun 26;10(1):131. doi: 10.1186/s13045-017-0491-2. PMID 28651604

RESULTS

PARTICIPANT FLOW:
Groups:
- Lenalidomide: The protocol initially employed a syncopated dosage regimen in which 10 mg of lenalidomide was taken orally once daily on Days 1 to 21 of a 28-day cycle, but was subsequently amended to employ a continuous dosage regimen in which 10 mg of lenalidomide was taken without a planned rest period. Participants who initially began therapy on the syncopated regimen and who did not experience dose-limiting adverse events (AEs) were allowed to switch to the continuous regimen.
Period: Overall Study
Arm/Group | Lenalidomide
Started | 148
Modified Intent to Treat Population | 94
Completed | 24 (24 patients rolled over to free drug due to sponsor closure of study.)
Not Completed | 124
Not completed — Adverse Event | 37
Not completed — Lack of Efficacy | 52
Not completed — Withdrawal by Subject | 8
Not completed — Lost to Follow-up | 1
Not completed — Death | 11
Not completed — Study Closed by Sponsor | 2
Not completed — Disease Progression | 7
Not completed — Investigator Decision | 2
Not completed — Non-Compliance | 2
Not completed — Loss of Response | 1
Not completed — Secondary Malign Disease | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide
Number analyzed (Participants) | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (10.50)
Age, Customized [Number; unit: participants]
  <= 65 years | 48
  >65 years | 100
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97
  Male | 51
Race/Ethnicity, Customized [Number; unit: participants]
  White | 143
  Hispanic | 3
  Asian/Pacific Islander | 2
Region of Enrollment [Number; unit: participants]
  United States | 112
  Germany | 36
Duration of Myelodysplastic Syndrome (MDS) [Mean (Standard Deviation); unit: years] — Time from diagnosis of MDS until study start.
  years | 3.4 (3.29)
Participants with 5q(-) (31-33) Chromosomal Abnormality [Number; unit: participants] | 148
International Prognostic Scoring System (IPSS) Score [Number; unit: participants] — The international prognostic scoring system (IPSS) is a standard for risk assessment in primary myelodysplastic syndromes (MDS) that categorizes prognoses taking into account cytogenetics, cytopenias, blasts and blood counts. The IPSS prognostic subgroups consist of low-, intermediate-1-, intermediate-2-, and high-risk groups. The scale is 0-3.5 at 0.5 increments. Scores of 0=Low; 0.5-1.0=Int-1; 1.5-2.0=Int-2; 2.5-3.5=High risk which corresponds to poorer prognosis. The assessment was performed by the Central Reviewer.
  participants
    Low (0) | 49
    Intermediate-1 (0.5 to 1.0) | 69
    Intermediate-2 (1.5 to 2.0) | 7
    High (>=2.5) | 2
    Missing (unable to assign) | 21
French-American-British (FAB) Classification [Number; unit: participants] — FAB is a classification system for five (5) subtypes of myelodysplastic syndrome that are distinguished by the percentage of myeloblasts, presence or absence of ringed sideroblasts or a monocytosis. Classification was made by the Central Reviewer.
  participants
    Refractory anemia (RA) | 78
    Refractory anemia with ringed sideroblasts (RARS) | 16
    Refractory anemia with excess blasts (RAEB) | 30
    Chronic myelomonocytic leukemia (CMML) | 3
    Acute leukemia | 1
    Unable to classify | 20
Cytogenetic Complexity [Number; unit: participants]
  Isolated 5q | 110
  Intermediate (5q + 1 abnormality) | 25
  Complex | 12
  Unknown | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — ECOG indicates a person's ability to perform life's functions on a scale of 0-5:
  0= fully active and no restrictions
  1. restricted but ambulatory and capable of light work
  2. ambulatory and capable of self-care but unable to work
  3-4= increasingly restricted
  5= dead
  participants
    0 | 59
    1 | 75
    2 | 14
    3 - 5 | 0

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Achieved Red Blood Cell (RBC) -Transfusion Independence
Description: Number of participants who achieved RBC-transfusion independence, which was defined as the absence of an intravenous infusion of any RBC transfusion during any consecutive "rolling" 56 days during the treatment period (eg, Days 1 to 56, Days 2 to 57, Days 3 to 58, etc), and accompanied by at least a 1 g/dL increase from screening/baseline in hemoglobin.
Time Frame: Up to 2 years
Population: Modified Intent to Treat (MITT)
  * diagnosis of low- or int-1-risk MDS associated with a del(5q) cytogenetic abnormality based on central hematologic and cytogenetic reviewers confirmation
  * received ≥2 transfusions in each of the 8-week periods during the 16 week pre-treatment period
  * received ≥1 dose of study drug
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 94
participants | 59

2. Secondary Outcome: Participants With Adverse Experiences
Description: Counts of study participants who had adverse events (AEs) during the study. A participant with multiple occurrences of an adverse event within a category is counted only once in that category. Adverse events were evaluated by the investigator.
  The National Cancer Institute (NCI)'s Common Toxicity Criteria for AEs (NCI CTC) was used to grade AE severity. Severity grade 3= severe and undesirable AE. Severity grade 4= life-threatening or disabling AE.
Time Frame: Up to 2 Years
Population: Safety population included all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 148
participants
  At least one AE | 148
  At least one AE related to study drug | 143
  At least one NCI CTC grade 3-4 AE | 140
  At least one NCI CTC grade 3-4 AE related to drug | 131
  At least one serious AE | 89
  At least one serious AE related to study drug | 40
  AE leading to dose reduction or interruption | 131
  AE leading to discontinuation of study drug | 47

3. Secondary Outcome: Participants With a >= 50% Decrease From Baseline in Red Blood Cell (RBC) Transfusion Requirements Over Any Consecutive 56 Days During Study
Description: A participant was categorized as having a transfusion reduction response if there was a ≥ 50% decrease from pretreatment transfusion requirements (before the start of the study mediation) compared to any consecutive 56 days during the study (i.e. post treatment).
Time Frame: Baseline (Day -54 to Day 0), During study (Day 1 up to 2 years)
Population: as for outcome 1
Measure: Number; unit: participant
Arm/Group | Lenalidomide
Number analyzed (Participants) | 94
participant | 70

4. Secondary Outcome: Time to Transfusion Independence
Description: Transfusion independence was defined as the absence of an intravenous infusion of any RBC transfusion during any consecutive "rolling" 56 days during the treatment period (e.g., Days 1 to 56, Days 2 to 57, Days 3 to 58, etc.), and accompanied by at least a 1 g/dL increase from screening/baseline in hemoglobin. Time to transfusion independence was defined as the day of the first dose of study drug to the first day of the first 56-day RBC transfusion-free period.
Time Frame: up to 2 years
Population: Modified intent to treat population who achieved transfusion independence
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Lenalidomide
Number analyzed (Participants) | 59
weeks | 6.2 (6.89)

5. Secondary Outcome: Participants Who Relapsed or Maintained Their Transfusion Independence After Achieving Transfusion Independence During the Study
Description: Transfusion independence was defined as the absence of an intravenous infusion of any RBC transfusion during any consecutive "rolling" 56 days during the treatment period (e.g., Days 1 to 56, Days 2 to 57, Days 3 to 58, etc.), and accompanied by at least a 1 g/dL increase from screening/baseline in hemoglobin. Participants who relapsed required a transfusion after the period of transfusion independence. Participants who maintained transfusion independence did not require a transfusion during the remainder of the study.
Time Frame: up to 2 years
Population: Modified intent to treat population who achieved transfusion independence
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 59
participants
  Relapsed (had a transfusion after response) | 35
  Maintained transfusion independence | 24

6. Secondary Outcome: Kaplan Meier Estimate for Duration of Transfusion Independence Response
Description: Duration of response is measured from the first of the consecutive 56 days during which the participant was free of RBC transfusions to the date of the first RBC transfusion after this period. Duration of response was censored at the date of last visit for participants who maintained transfusion independence.
Time Frame: up to 2 years
Population: Modified intent to treat population who achieved transfusion independence
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenalidomide
Number analyzed (Participants) | 59
weeks | 97.0 [52.9 to 191.9]

7. Secondary Outcome: Change in Hemoglobin Concentration From Baseline to Maximum Value During Response Period for Responders
Description: The change from baseline in hemoglobin for participants who became RBC-transfusion independent. The maximum hemoglobin value obtained during the response period is used in the calculation of change from baseline.
Time Frame: Baseline (Day -54 to Day 0), During study (Day 1 up to 2 years)
Population: Modified intent to treat population who achieved transfusion independence
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Lenalidomide
Number analyzed (Participants) | 59
g/dL | 6.1 (1.92)

8. Secondary Outcome: Participant Counts of Cytogenetic Response
Description: Participants deemed evaluable by the central cytogenetic review had their cytogenetic response categorized as major or minor. A major cytogenetic response was defined as ≥ 20 metaphases recorded at baseline, and at least
  1 post baseline evaluation with ≥ 20 metaphases analyzed with no abnormal metaphases observed. A minor cytogenetic response was defined as ≥ 20 metaphases analyzed at baseline, and at least 1 post baseline evaluation with ≥ 20 metaphases analyzed with a ≥ 50% reduction in the proportion of hematopoietic cells with cytogenetic abnormalities compared with baseline.
Time Frame: up to 2 years
Population: Evaluable participants from the modified intent to treat population. Evaluable participants had ≥ 20 metaphases analyzed at baseline during the 56-day period immediately preceding the first day of study drug intake and ≥ 20 metaphases analyzed at least once at postbaseline visits.
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 52
participants
  Major | 18
  Minor | 20
  None | 14

9. Secondary Outcome: Participant Counts of Platelet Response
Description: Major platelet response: participants with a minimum pretreatment platelet of <100,000/mm^3 in all values within 56 days of start of treatment, an absolute increase of ≥30,000/mm^3 sustained for ≥56 consecutive days. In platelet transfusion-dependent participants, a major response was stabilization of platelet counts and platelet transfusion independence.
  Minor platelet response: participants with a minimum pretreatment platelet of <100,000/mm^3, a ≥ 50% increase in platelet count with a net increase >10,000/mm^3 for a consecutive 56-day period in the absence of platelet transfusions.
Time Frame: up to 2 years
Population: Evaluable participants from the modified intent to treat population. Participants must have a baseline platelet count <100 * 10^9/L to be included in the analysis.
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 15
participants
  Major | 2
  Minor | 0
  None | 13

10. Secondary Outcome: Participant Counts of Absolute Neutrophil Count (ANC) Response
Description: Major neutrophil response: participants with a minimum pretreatment ANC concentration of < 1500/mm^3 in all values obtained within 56 days of start of treatment, a ≥ 100% increase or an absolute increase of
  ≥ 500/mm^3, whichever was greater (at least to be ≥ 500/mm^3), sustained for 56 consecutive days. Minor neutrophil response: participants with a minimum pretreatment ANC concentration of < 1500/mm^3, an increase in ANC concentration of ≥ 100% sustained for 56 consecutive days.
Time Frame: up to 2 years
Population: Evaluable participants from the modified intent to treat population. Evaluable participants are required to have a baseline absolute neutrophil count (ANC) <1 * 10^9/L.
Measure: Number; unit: participant
Arm/Group | Lenalidomide
Number analyzed (Participants) | 27
participant
  Major | 9
  Minor | 0
  None | 18

11. Secondary Outcome: Participants With Complete or Partial Bone Marrow Improvement
Description: Bone marrow aspirates were assessed by a central reviewer. A complete bone marrow improvement required a baseline French-American-British (FAB) classification (see Baseline Characteristics) of refractory anemia (RA), refractory anemia with ringed sideroblasts (RARS), refractory anemia with excess blasts (RAEB) or chronic myelomonocytic leukemia (CMML) and a during study assessment of no MDS. A partial bone marrow improvement reflected an improved FAB classification compared to baseline (e.g. RARS to RA) but evidence of MDS continued to exist.
Time Frame: up to 2 years
Population: Modified intent to treat population of participants with adequate bone marrow aspirate at baseline.
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 94
participants
  Complete bone marrow improvement | 22
  Partial bone marrow improvement | 15

12. Secondary Outcome: Participants With Bone Marrow Progression
Description: Bone marrow aspirate was assessed by a central reviewer. Progression is represented in two categories according to changes from baseline in French-American-British (FAB) classification (see Baseline Characteristics):
  * Baseline classification of refractory anemia (RA) or refractory anemia with ringed sideroblasts (RARS) to a during treatment (plus 30 days) classification of refractory anemia with excess blasts (RAEB).
  * Any baseline FAB classification to a during treatment (plus 30 days) classification of acute myeloid leukemia (AML).
Time Frame: up to 2 years
Population: Modified intent to treat population of participants with adequate bone marrow aspirate at baseline.
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 94
participants
  RA/RARS to RAEB | 11
  RA/RARS/RAEB/CMML to AML | 6

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Lenalidomide
Serious Adverse Events (participants affected / at risk) | 89/148
Other Adverse Events (participants affected / at risk) | 148/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=148)
Pneumonia Not Otherwise Specified (NOS) (Infections and infestations) | 15
Neutropenia (Blood and lymphatic system disorders) | 10
Anaemia NOS (Blood and lymphatic system disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 8
Febrile Neutropenia (Blood and lymphatic system disorders) | 8
Acute Leukaemia NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Cardiac Failure Congestive (Cardiac disorders) | 6
Sepsis NOS (Infections and infestations) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Deep Vein Thrombosis (Vascular disorders) | 5
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 5
Vomiting NOS (Gastrointestinal disorders) | 5
Abdominal Pain NOS (Gastrointestinal disorders) | 4
Diarrhoea NOS (Gastrointestinal disorders) | 4
Pyrexia (General disorders) | 4
Acute Myeloid Leukaemia NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Atrial Fibrillation (Cardiac disorders) | 3
Dizziness (Nervous system disorders) | 3
Gastroenteritis NOS (Gastrointestinal disorders) | 3
Leukopenia NOS (Blood and lymphatic system disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Pancytopenia (Blood and lymphatic system disorders) | 3
Asthenia (General disorders) | 2
Bacteraemia (Infections and infestations) | 2
Cardiac Failure NOS (Cardiac disorders) | 2
Cellulitis (Infections and infestations) | 2
Cerebrovascular Accident (Nervous system disorders) | 2
Depressed Level of Consciousness (Nervous system disorders) | 2
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 2
Fall (General disorders) | 2
Fatigue (General disorders) | 2
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 2
Femur Fracture (Injury, poisoning and procedural complications) | 2
Infection NOS (Infections and infestations) | 2
Medical Device Complication (Injury, poisoning and procedural complications) | 2
Multi-Organ Failure (General disorders) | 2
Myocardial Infarction (Cardiac disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Hypertension NOS (Respiratory, thoracic and mediastinal disorders) | 2
Rash NOS (Skin and subcutaneous tissue disorders) | 2
Rectal Haemorrhage (Gastrointestinal disorders) | 2
Renal Failure NOS (Renal and urinary disorders) | 2
Syncope (Nervous system disorders) | 2
Transient Ischaemic Attack (Nervous system disorders) | 2
Urinary Tract Infection NOS (Infections and infestations) | 2
Acute Febrile Neutrophilic Dermatosis (Skin and subcutaneous tissue disorders) | 1
Aphasia (Nervous system disorders) | 1
Arthrlagia (Musculoskeletal and connective tissue disorders) | 1
Asthma NOS (Respiratory, thoracic and mediastinal disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
B-Cell Lymphoma NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Blood Creatinine Increased (Investigations) | 1
Bronchitis Acute NOS (Infections and infestations) | 1
Carcinoid Tumour of the Small Bowel (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cardio-Respiratory Arrest (Cardiac disorders) | 1
Cardiomyopathy NOS (Cardiac disorders) | 1
Central Line Infection (Infections and infestations) | 1
Cerebral Haemorrhage (Nervous system disorders) | 1
Cervical Dysplasia (Reproductive system and breast disorders) | 1
Chest Pain (General disorders) | 1
Cholecystitis NOS (Hepatobiliary disorders) | 1
Chronic Obstructive Airways Disease Exacerbated (Respiratory, thoracic and mediastinal disorders) | 1
Clostridial Infection NOS (Infections and infestations) | 1
Coagulopathy (Blood and lymphatic system disorders) | 1
Colitis Ischaemic (Gastrointestinal disorders) | 1
Colonic Polyp (Gastrointestinal disorders) | 1
Comminuted Fracture (Injury, poisoning and procedural complications) | 1
Constipation (Gastrointestinal disorders) | 1
Convulsions NOS (Nervous system disorders) | 1
Dementia NOS (Nervous system disorders) | 1
Dermatitis Medicamentosa (Skin and subcutaneous tissue disorders) | 1
Diastolic Dysfunction (Cardiac disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Enterobacter Sepsis (Infections and infestations) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Gastritis NOS (Gastrointestinal disorders) | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1
Groin Infection (Infections and infestations) | 1
Headache (Nervous system disorders) | 1
Herpes Zoster (Infections and infestations) | 1
Hiatus Hernia (Gastrointestinal disorders) | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypersensitivity NOS (Immune system disorders) | 1
Hypertensive Encephalopathy (Nervous system disorders) | 1
Hypoglycaemia NOS (Metabolism and nutrition disorders) | 1
Hypotension NOS (Vascular disorders) | 1
Influenza (Infections and infestations) | 1
Intermittent Pyrexia (General disorders) | 1
Intestinal Perforation NOS (Gastrointestinal disorders) | 1
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1
Klebsiella Sepsis (Infections and infestations) | 1
Lobar Pneumonia NOS (Infections and infestations) | 1
Localised Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Infiltration NOS (Respiratory, thoracic and mediastinal disorders) | 1
Migraine NOS (Nervous system disorders) | 1
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal Perforation (Gastrointestinal disorders) | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 1
Ovarian Cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Overdose NOS (Injury, poisoning and procedural complications) | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Peripheral Ischaemia (Vascular disorders) | 1
Perirectal Abscess (Gastrointestinal disorders) | 1
Post Procedural Site Wound Infection (Infections and infestations) | 1
Pulmonary Oedema NOS (Cardiac disorders) | 1
Refractory Anaemia with Excess Blasts in Transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal Failure Acute (Renal and urinary disorders) | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Rigors (General disorders) | 1
Senile Dementia NOS (Nervous system disorders) | 1
Sinusitis Acute NOS (Infections and infestations) | 1
Sinusitis NOS (Infections and infestations) | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1
Subarachnoid Haemorrhage NOS (Nervous system disorders) | 1
Subdural Haematoma (Nervous system disorders) | 1
Sudden Death (General disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Thrombophlebitis Superficial (Vascular disorders) | 1
Thymoma NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Troponin I Increased (Investigations) | 1
Vaginosis Fungal NOS (Infections and infestations) | 1
Vertigo (Ear and labyrinth disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=148)
Thrombocytopenia (Blood and lymphatic system disorders) | 93
Neutropenia (Blood and lymphatic system disorders) | 91
Diarrhoea Not Otherwise Specified (NOS) (Gastrointestinal disorders) | 87
Pruritus (Skin and subcutaneous tissue disorders) | 66
Fatigue (General disorders) | 62
Rash NOS (Skin and subcutaneous tissue disorders) | 54
Arthralgia (Musculoskeletal and connective tissue disorders) | 46
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 44
Nausea (Gastrointestinal disorders) | 41
Oedema Peripheral (General disorders) | 40
Back Pain (Musculoskeletal and connective tissue disorders) | 39
Constipation (Gastrointestinal disorders) | 39
Cough (Respiratory, thoracic and mediastinal disorders) | 38
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 37
Pyrexia (General disorders) | 37
Dizziness (Nervous system disorders) | 35
Headache (Nervous system disorders) | 33
Upper Respiratory Tract Infection NOS (Infections and infestations) | 33
Anaemia NOS (Blood and lymphatic system disorders) | 32
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 31
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 29
Pain in Limb (Musculoskeletal and connective tissue disorders) | 25
Abdominal Pain NOS (Gastrointestinal disorders) | 24
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 24
Asthenia (General disorders) | 22
Hypokalaemia (Metabolism and nutrition disorders) | 22
Dry Skin (Skin and subcutaneous tissue disorders) | 21
Urinary Tract Infection NOS (Infections and infestations) | 21
Anorexia (Metabolism and nutrition disorders) | 20
Insomnia (Psychiatric disorders) | 19
Leukopenia NOS (Blood and lymphatic system disorders) | 19
Myalgia (Musculoskeletal and connective tissue disorders) | 19
Sinusitis NOS (Infections and infestations) | 19
Contusion (Skin and subcutaneous tissue disorders) | 18
Oedema NOS (General disorders) | 18
Vomiting NOS (Gastrointestinal disorders) | 18
Bronchitis NOS (Respiratory, thoracic and mediastinal disorders) | 17
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 16
Night Sweats (Skin and subcutaneous tissue disorders) | 16
Abdominal Pain Upper (Gastrointestinal disorders) | 14
Acquired Hypothyroidism (Endocrine disorders) | 14
Depression (Psychiatric disorders) | 14
Pain NOS (General disorders) | 14
Peripheral Swelling (Musculoskeletal and connective tissue disorders) | 14
Fall (General disorders) | 13
Hypertension NOS (Vascular disorders) | 13
Sweating Increased (Skin and subcutaneous tissue disorders) | 13
Alanine Aminotransferase Increased (Investigations) | 12
Cellulitis (Infections and infestations) | 12
Dry Mouth (Gastrointestinal disorders) | 12
Dysuria (Renal and urinary disorders) | 12
Erythema (Skin and subcutaneous tissue disorders) | 12
Loose Stools (Gastrointestinal disorders) | 12
Rhinitis NOS (Respiratory, thoracic and mediastinal disorders) | 12
Weight Decreased (Investigations) | 12
Chest Pain (General disorders) | 11
Hypoaesthesia (Nervous system disorders) | 11
Hypomagnesaemia (Metabolism and nutrition disorders) | 11
Influenza (Infections and infestations) | 11
Toothache (Gastrointestinal disorders) | 11
Alopecia (Skin and subcutaneous tissue disorders) | 10
Dysgeusia (Nervous system disorders) | 10
Ecchymosis (Skin and subcutaneous tissue disorders) | 10
Pain in Foot (Musculoskeletal and connective tissue disorders) | 10
Palpitations (Cardiac disorders) | 10
Paraesthesia (Nervous system disorders) | 10
Peripheral Neuropathy NOS (Nervous system disorders) | 10
Conjunctivitis (Eye disorders) | 9
Rigors (General disorders) | 9
Anxiety (Psychiatric disorders) | 8
Appetite Decreased NOS (Metabolism and nutrition disorders) | 8
Flatulence (Gastrointestinal disorders) | 8
Herpes Simplex (Infections and infestations) | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 8
Neck Pain (Musculoskeletal and connective tissue disorders) | 8
Peripheral Sensory Neuropathy (Nervous system disorders) | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8
Skin Lesions NOS (Skin and subcutaneous tissue disorders) | 8
Vision Blurred (Eye disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Unless approved by Celgene, single center data will not be published before multicenter data, unless more than 1 year has elapsed since completion of the Study. Thereafter, Investigator may publish single center data provided that Investigator shall: i) provide a copy of the publication to Celgene at least 60 days in advance of submission for publication; ii) delete Celgene Confidential Information and; iii) delay submission up to 90 additional days to permit intellectual property filings.